CLINICAL TRIAL: NCT06530368
Title: Investigation of the Effect of a Calisthenic Home Exercise Program on Premenstrual Symptoms, Pain and Sleep Quality in Young Women
Brief Title: Effect of a Calisthenic Exercises on Premenstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, PT, MSc., Halic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28.07.2024-MÇ
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Control group (No Intervention): Participants in the first group were not subjected to any intervention and were asked not to participate in any exercise program for eight weeks.
- Group 2: Calisthenic home exercise group (Experimental): Participants in the second group were informed about calisthenic home exercise programs face to face and were asked to perform these exercises as home exercises for eight weeks.
  Interventions: Other: Calisthenic home exercise programs

INTERVENTIONS:
Other: Calisthenic home exercise programs — Participants in the second group were informed about calisthenic home exercise programs face to face and were asked to perform these exercises as home exercises for eight weeks.
  Arms: Group 2: Calisthenic home exercise group

SUMMARY:
The aim of this study is to examine the effects of an eight-week calisthenic home exercise program on premenstrual symptoms, pain and sleep quality in young women.

DETAILED DESCRIPTION:
The study was conducted on 30 volunteers who met the inclusion criteria among female students studying at Haliç University Faculty of Health Sciences. The "Premenstrual Syndrome Scale (PMSS)" was used to assess the individuals' premenstrual symptoms; the "Visual Analog Scale (VAS)" was used to assess pain for each of the abdominal, lumbar and general body pain; and the "Pittsburgh Sleep Quality Index (PSQI)" was used to assess sleep quality. Then, the participants were randomly divided into two groups as "Group 1: Control group (n=15)" and "Group 2: - Calisthenic home exercise group (n=15)". Participants in the first group were not subjected to any intervention and were asked not to participate in any exercise program for eight weeks. Participants in the second group were informed about calisthenic home exercise programs face to face and were asked to perform these exercises as home exercises for eight weeks. At the end of the treatment process, participants' PMSS, VAS and PSQI scores were re-evaluated.Statistical analysis will be performed with SPSS 24.0 program. If the data is parametric, paired sample t-test will be used for within-group evaluation; independent sample t-test will be used for between-group evaluation. If the data is non-parametric, Wilson test will be used for within-group evaluation and Mann Whitney U test will be used for between-group evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18-25
* Studying at Halic University Faculty of Health Sciences
* Voluntarily participating in the study
* Having a normal menstrual cycle
* Not exercising
* Having a score above the mild level on the Premenstrual Syndrome Scale

Exclusion Criteria:

* Having a condition that prevents exercise
* Pregnancy
* Menopause
* Having a gynecological disease (endometriosis, ovarian cyst, pelvic infection, myoma/uterine tumor, etc.)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women
Enrollment: 30 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | at baseline and at week 8.
  The scale, which is widely used in the clinic, has 44 questions that women mark considering "the state of being in the period one week before menstruation". The lowest score that can be obtained from the scale is 44; the highest score is 220. In addition, PMS severity classes can be created according to the scores obtained from the scale. Accordingly, a score of 88 and above from PMSS indicates severe PMS symptoms, and a score below 88 indicates mild PMS symptoms. Individuals who scored 88 and above from the scale were included in our study.
Visual Analog Scale (VAS) | at baseline and at week 8.
  VAS is a simple, practical, valid, reliable and repeatable measure that evaluates the pain felt by scoring it between 0-10. Participants were asked to score the pain intensity they felt between 0-10 for each of the abdominal region, lumbar region and general body pain.
Pittsburgh Sleep Quality Index (PSQI) | at baseline and at week 8.
  The PSQI questionnaire used to assess sleep quality includes 18 items for scoring. A total PSQI score between 0-4 indicates good sleep quality, and a score between 5-21 indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Şahin Altaç, PT, MSc., Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pearce E, Jolly K, Jones LL, Matthewman G, Zanganeh M, Daley A. Exercise for premenstrual syndrome: a systematic review and meta-analysis of randomised controlled trials. BJGP Open. 2020 Aug 25;4(3):bjgpopen20X101032. doi: 10.3399/bjgpopen20X101032. Print 2020 Aug. PMID 32522750
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Mohebbi Dehnavi Z, Jafarnejad F, Sadeghi Goghary S. The effect of 8 weeks aerobic exercise on severity of physical symptoms of premenstrual syndrome: a clinical trial study. BMC Womens Health. 2018 May 31;18(1):80. doi: 10.1186/s12905-018-0565-5. PMID 29855308